CLINICAL TRIAL: NCT03726060
Title: Effectiveness of Physical Teraphy in the Treatment of Myogenic Temporomandibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paolo Pillastrini (Other)
Responsible Party: Sponsor-Investigator, Paolo Pillastrini, professor, University of Bologna
Organization: University of Bologna (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 47/2018/SPER/AUSLBO
Record Dates: First submitted 2018-10-24; First posted 2018-10-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Control Groups; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- splint therapy (Other): Alginate impressions will be taken and the plaster models of the dental arches will be made.
  The splint will be subsequently delivered to the patient with the relative indications of use.
  The splint therapy consist in the use of neuromuscoral splint every the night for 6 months.
  Interventions: Other: control group
- physical therapy with splint therapy (Other): The treatment consists of a series of interventions: advice on self-treatment techniques to be performed at home and administering manual therapy techniques addressed to: temporomandibular district, cervical and cervico-thoracic junction.
  Each session will be carried out individually and will last for 45 minutes. This duration will be divided as follows: 25 minutes dedicated to the temporomandibular district, 15 minutes to the cervical and cervico-thoracic junction, 5 minutes to teaching self-treatment techniques to be carried out at home and to verify the correct way of performing them.
  The cycle will consist of 10 sessions distributed over 3 months.
  Interventions: Other: test group

INTERVENTIONS:
Other: control group — In the control group the patient will undergo gnathologic therapy for 6 months with neuromuscural splint every night for 3 months
  Other Names: splint therapy
  Arms: splint therapy
Other: test group — In the test group the patient will undergo gnathologic therapy with neuromuscural splint every night for 3 months in association with physical therapy
  Other Names: splint therapy with physical therapy
  Arms: physical therapy with splint therapy

SUMMARY:
The aim of study is evaluate the effectiveness of physical therapy in of the treatment myogenic temporomandibular disorders.

They will enrolled 100 patient which will be divided into two groups. The primary objective is evaluate the effectiveness of physiotherapy on pain (measured with the Visual Analogic Scale - VAS scale).

The second objective is evaluate mandibular motion (by measuring the range of motion - ROM) and investigate the presence of psychosocial factors (using the Anxiety and Depression Scale - HADS questionnaire).

DETAILED DESCRIPTION:
Randomized controlled clinical trial with randomization according to a multi-phase design.

Phase 1 involves the enrollment of patients with DTMs based on diagnostic criteria.

Phase 2 includes the algogenic, kinetic and gnathological evaluation of the enrolled patients.

Phase 3 provides for the adoption of the criterion to one of the 2 treatment groups on the basis of the randomization list.

The 2 therapeutic protocols are:

* gnathological therapy (splint) associated with education and physiotherapy (test group);
* gnathological therapy (splint) associated with education (control group). During the first visit the patient will be enlisted by evaluating the inclusion and exclusion criteria and signed the informed consent, he / she will be assigned a unique identification code.

The code consists of a progressive number followed by the patient's initials (eg 01-F.R.).

Subsequently, the patients will be randomized blinded and assigned to one of the two study groups.

Randomization will be performed using random, computer-generated, centralized numbers placed in sealed opaque envelopes provided by the study coordinator.

Both types of treatment will be performed by a single operator respectively.

ELIGIBILITY:
Inclusion Criteria:

* patients with myogenic temporomandibular disorders assessed with clinical examination as established by the DC / TMD1;
* patients older than 18 years;
* good knowledge of Italian language;
* patients who have signed informed consent

Exclusion Criteria:

* edentulism which makes it impossible to apply gnathological bite;
* patients with psychiatric problems;
* patients included in other experimental protocols;
* patients already undergoing surgical and / or radial therapy of the cervical and facial areas;
* other temporomandibular disorders without a myogenic component;
* treatment of the cervical and TMJ district in the previous 3 months;
* history of drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of physical therapy using the VAS scale which allows to measure the varation of pain | Change from initial VAS at 3 and 6 months from the beginning of the treatment
  The VAS measures the intensity of the pain that thethe patient perceived and it is represented by a 10 cm long scale with a score from 0 to 10. The VAS will be evaluated in 3 times: at rest; during the maximum buccal opening; during chewing

SECONDARY OUTCOMES:
ROM (range of motion) | The measurement of the ROM occurs at the recruitment then at 3 and 6 months from the beginning of the treatment
  The ROM measures the joint function. It provides the analytical and millimetric measurement of functional movements with a precision gauge positioned between the incisal edges of the upper and lower anterior groups.
  It should be noted: maximum buccal opening; deviation of the median line; left and right lateral movements; overjet and overbite.
  It should also be noted the extent of final elasticity (or end-feel test and its nature (elastic, painful, hard)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bologna, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Romeo A, Incorvati C, Vanti C, Turolla A, Marinelli F, Defila L, Gulotta C, Marchetti C, Pillastrini P. Physical therapy in addition to occlusal splint in myogenic temporomandibular disorders: A randomised controlled trial. J Oral Rehabil. 2024 Aug;51(8):1566-1578. doi: 10.1111/joor.13729. Epub 2024 May 17. PMID 38757854
- [Derived] Incorvati C, Romeo A, Fabrizi A, Defila L, Vanti C, Gatto MRA, Marchetti C, Pillastrini P. Effectiveness of physical therapy in addition to occlusal splint in myogenic temporomandibular disorders: protocol of a randomised controlled trial. BMJ Open. 2020 Aug 13;10(8):e038438. doi: 10.1136/bmjopen-2020-038438. PMID 32792449